CLINICAL TRIAL: NCT05236491
Title: COvid-19 Vaccine Booster in Immunocompromised Rheumatic Diseases
Acronym: COVBIRD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul R Fortin (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Paul R Fortin, Rheumatologist, Clinical Researcher, Principal Investigator, CHU de Quebec-Universite Laval
Organization: CHU de Quebec-Universite Laval (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COVB-2022-1
Record Dates: First submitted 2022-02-10; First posted 2022-02-11 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis; Autoimmune Rheumatologic Disease; Systemic Lupus Erythematosus; Systemic Vasculitis; Systemic Sclerosis; Scleroderma; Undifferentiated Connective Tissue Diseases; Overlap Connective Tissue Disease; Immunosuppression
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Systemic Vasculitis; Scleroderma, Systemic; Scleroderma, Diffuse; Undifferentiated Connective Tissue Diseases; MASS syndrome | interventions — COVID-19 Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Trajectory A (Active Comparator): Participants who have received 3 doses of an mRNA vaccine, will be offered a choice between a fourth dose of an mRNA vaccine and a dose of a protein subunit vaccine (PSV) (Novavax NUVAXOVID)
  For the Moderna SPIKEVAX Bivalent Original/Omicron BA.4/5: participants will receive one (1) intramuscular injection of 0.5 mL (50 mcg).
  For the Novavax Nuvaxovid vaccine: participants will receive one (1) intramuscular injection of 0.5 mL (5 mcg) of Novavax Nuvaxovid.
  Interventions: Biological: COVID-19 vaccine
- Trajectory B (No Intervention): Participants who have already received a 4 doses or more of COVID-19 vaccine in the community at inclusion and do not wish to receive a 5th dose of vaccine in the study.
- Trajectory B5 (Active Comparator): Participants who have received 4 doses of an mRNA vaccine at inclusion and wish to receive a dose of a protein subunit vaccine (PSV) (Novavax NUVAXOVID) as a fifth dose.
  For the Novavax Nuvaxovid vaccine: participants will receive one (1) intramuscular injection of 0.5 mL (5 mcg) of Novavax Nuvaxovid.
  Interventions: Biological: COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine — Participants are to receive a booster dose of a COVID-19 vaccine.
  Arms: Trajectory A; Trajectory B5

SUMMARY:
People living with Systemic autoimmune rheumatic diseases (SARDs) face a new and urgent dilemma: immunosuppression increases risk for worse COVID-19 infection, yet an immune stimulation, such as vaccination, could re-activate their disease. Fear of vaccine-related disease reactivation is not of concern in other immunosuppressed groups (e.g. patients receiving chemotherapy or hemodialysis) but in SARDs, disease flare could lead to organ failure or even death. Specific research in this population is therefore critical. Moreover, among SARD patients, those on anti-CD-20 monoclonal antibody (mAb) (i.e. rituximab (anti-CD-20 mAb)), a medication used to treat inflammatory types of arthritis, have extremely low immunity post-COVID-19 mRNA vaccine. This study will test the hypothesis that a booster dose of a COVID-19 vaccine is safe and enhances post-vaccine humoral and cellular responses in SARDs patients on anti-CD-20 mAb treatment. The magnitude of this response depends on the type of COVID-19 vaccine administered and is optimal when the booster dose is a vaccine from a different group than the one used for primary immunization (mix-and-match approach).

DETAILED DESCRIPTION:
Systemic autoimmune rheumatic diseases (SARDs) include rheumatoid arthritis (RA), systemic lupus (SLE), systemic vasculitis, and related diseases where immune system activity causes widespread inflammation in organs, leading to sickness, organ damage, disability, high health costs, and even death. With no cure, SARDs require life-long immunosuppression. People living with SARDs now face a new and urgent dilemma: immunosuppression increases risk for worse COVID-19 infection, yet an immune stimulation, such as vaccination, could re-activate their disease. Fear of vaccine-related disease reactivation is not of concern in other immunosuppressed groups (e.g. patients receiving chemotherapy or hemodialysis) but in SARDs, disease flare could lead to organ failure or even death. Specific research in this population is therefore critical. Moreover, among SARD patients, those on anti-CD-20 monoclonal antibody (mAb) (i.e. rituximab (anti-CD-20 mAb)) have extremely low humoral immunity post-COVID-19 mRNA vaccine. As of mid-July 2021, 1489 SARDs patients were actively treated with anti-CD-20 mAb in the province of Quebec (personal communication).

This study will test the hypothesis that a booster dose of a COVID-19 vaccine is safe and enhances post-vaccine humoral and cellular responses in SARDs patients on anti-CD-20 mAb treatment. The magnitude of this response depends on the type of COVID-19 vaccine administered and is optimal when the booster dose is a vaccine from a different group than the one used for primary immunization (mix-and-match approach).

Our goal is to recruit 287 adults with SARDs on anti-CD-20 mAb treatment post-three doses of an approved mRNA-COVID-19 vaccine in a non-randomized, open label, comparative clinical trial with pragmatic features. This includes persons with rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), systemic sclerosis (SSc), inflammatory immune myopathies (IIM), overlap and undifferentiated connective tissue diseases (OCTD and UCTD) and ANCA-associated vasculitis (AAV). We will test at entry all participants for their anti-SARS-CoV-2-spike receptor binding domain (anti-RBD) antibody response to their previous doses of mRNA-COVID-19 vaccines. For participants who have received 3 doses of an mRNA vaccine, we will offer them a choice between a fourth dose of an mRNA (vaccine and a dose of a protein subunit vaccine (PSV). For participants who have already received 4 doses of an mRNA vaccine in the community, they will be offered a dose of a protein subunit vaccine (PSV) as a fifth dose.

The primary study outcome will be the assessment of the safety and reactogenicity of a booster dose of COVID-19 vaccine using a mix-and-match strategy in immunocompromised rheumatic disease patients on an anti-CD-20 mAb. The secondary study outcome will be the humoral responses as measured by the anti-RBD Ab 28 days post vaccination. Exploratory outcomes include the cellular response at 28 days; the delayed humoral responses at 6 months; a comparison of the immunogenicity between types of vaccine (mRNA vs PSV); the evaluation of the effects of concomitant treatments on immunogenicity post-COVID-19 vaccine; the description of the rates of disease flares post booster dose of COVID-19 vaccine; and a description of the decision process for vaccine selection.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of a SARD (Rheumatoid arthritis, systemic lupus erythematosus (SLE), juvenile inflammatory arthritis, systemic sclerosis (SSc), idiopathic inflammatory myositis (IIM), overlap connective tissue diseases, mixed connective tissue disease, undifferentiated connective tissue diseases, giant-cell arteritis, and the ANCA-Associated Vasculitis: granulomatosis with polyangiitis (GPA; formerly known as Wegener's granulomatosis), microscopic polyangiitis (MPA), and eosinophilic granulomatosis with polyangiitis (EGPA; previously known as Churg-Strauss syndrome);
2. Has received 3 or more doses of an mRNA vaccine;
3. Age 18 years and older;
4. Male or non-pregnant female;
5. Rituximab treatment within last 12 months;
6. Able to comprehend the study protocol and provide informed consent.

Exclusion Criteria

1. Any medical disease or condition that, in the opinion of the site Principal Investigator or sub-investigator, precludes study participation;
2. Significant behavioral disturbances;
3. Previous diagnosis of hepatitis B, hepatitis C or HIV;
4. History of hypersensitivity or severe allergic reaction such as anaphylaxis to a component of the vaccine or to a previous vaccine;
5. People who experienced inflammation of the heart or lining of the heart (myocarditis or pericarditis) after a previous dose of an mRNA vaccine or protein subunit vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety of a booster dose of COVID-19 vaccine in patients on anti-CD-20 mAb. | 28 days
  Assessment of SARDs flares (self-reported and physician-confirmed) in relation to the time of the last dose of vaccine received. The frequency of 'significant flares' will be defined as worsening of RA symptoms (i.e., increase in DAS28 >1.2 or >0.6 if DAS28 at baseline was ≥3.2) with an increase in the number of swollen joints confirmed by a rheumatologist that is actionable (requires treatment intensification). For SLE, a flare will be defined as mild/moderate when the index SLEDAI increases by >3 and severe when it increases by >10. The need for treatment intensification (e.g., increase in the dose of steroids) will also be recorded as an indication of SLE flare. For AAV and other SARDs that do not have standard instruments to define flares, we will use the physician's assessment of the presence of a clinically significant flare to the general question " Has this patient experienced a clinically significant flare of their SARD? " and document relevant change in medication.
Reactogenicity of a booster dose of COVID-19 vaccine in patients on anti-CD-20 mAb. | 28 days
  Documentation of the reactogenicity to the booster dose of the vaccine. Reactogenicity post-booster dose will be based on the patient's diary and questionnaire collected at visit 28 days post booster dose vaccination.

SECONDARY OUTCOMES:
Humoral response | 28 days post vaccination
  We will define vaccine-induced humoral response as a positive (as defined by the cut-off of the assay) serum antibody response against the viral spike RBD protein 28 days post booster dose.
  We will measure 1)anti-RBD and anti-N antibodies in all participants at a minimum of three time points using the Héma-Québec assay (Dr Bazin) and 2)neutralization antibodies (NAbs) using the assay developed by Dr Flamand. In addition, we will use a panel of assays developed by Dr Finzi's group including assays to recognized variants of concern and antibody-dependent cell-mediated cytotoxicity (ADCC) and antibody-dependent cellular phagocytosis (ADCP) assays.

OTHER OUTCOMES:
Humoral response | 180 days post vaccination
  We will define vaccine-induced humoral response as a positive (as defined by the cut-off of the assay) serum antibody response against the viral spike RBD protein 28 days post booster dose.
  We will measure 1)anti-RBD and anti-N antibodies in all participants at a minimum of three time points using the Héma-Québec assay (Dr Bazin) and 2)neutralization antibodies (NAbs) using the assay developed by Dr Flamand. In addition, we will use a panel of assays developed by Dr Finzi's group including assays to recognized variants of concern and antibody-dependent cell-mediated cytotoxicity (ADCC) and antibody-dependent cellular phagocytosis (ADCP) assays.
Humoral response | 335 days post vaccination
  We will define vaccine-induced humoral response as a positive (as defined by the cut-off of the assay) serum antibody response against the viral spike RBD protein 28 days post booster dose.
  We will measure 1)anti-RBD and anti-N antibodies in all participants at a minimum of three time points using the Héma-Québec assay (Dr Bazin) and 2)neutralization antibodies (NAbs) using the assay developed by Dr Flamand. In addition, we will use a panel of assays developed by Dr Finzi's group including assays to recognized variants of concern and antibody-dependent cell-mediated cytotoxicity (ADCC) and antibody-dependent cellular phagocytosis (ADCP) assays.

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Fortin, MD,MPH,FRCPC, Principal Investigator — Centre de recherche du CHU de Québec - Université Laval
Locations (2):
- Canada (2):
  - Research Institute - McGill University Health Centre, Montreal, Quebec
  - Centre de recherche du CHU de Québec - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No